CLINICAL TRIAL: NCT06440525
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Impact of Intravenous RSLV-132 in Participants With Sjögren's Disease With Moderate to Severe Symptom Burden
Brief Title: A Study of RSLV-132 in Females With Sjögren's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Resolve Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 132-6
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Primary Sjögren Syndrome
MeSH Terms: interventions — RSLV-132

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- RSLV-132 (Experimental): Intravenous infusions of 10 mg/kg RSLV-132 solution on Days 1, 8, 15, 29, 43, 57, 71, 85, 99, 113, 127, 141, and 155) for a total of 22 weeks of treatment
  Interventions: Drug: RSLV-132
- Placebo (Placebo Comparator): Intravenous infusions of placebo solution on Days 1, 8, 15, 29, 43, 57, 71, 85, 99, 113, 127, 141, and 155) for a total of 22 weeks of treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RSLV-132 — Fc fusion protein comprised of catalytically active human ribonuclease (RNase) fused to human immunoglobulin G1 (IgG1)
  Arms: RSLV-132
Drug: Placebo — 0.9% sodium chloride solution
  Arms: Placebo

SUMMARY:
The goal of this clinical study is to learn if RSLV-132 improves the symptoms of SS in adults. It will also learn about the safety of RSLV-132. The main questions it aims to answer are:

* Does RSLV-132 improve the cardinal symptoms of Sjogren's including fatigue, dryness and pain?
* Does RSLV-132 improve the tiredness/fatigue caused by Sjogren's?
* What are the blood levels of RSLV-132 over time?
* What is the immune (antibody) response in the body to RSLV-132?
* What is the safety profile of RSLV-132?

Researchers will compare RSLV-132 to a placebo (a look-alike substance that contains no drug) to see if RSLV-132 improves the symptoms of pSS.

Participants will:

Take RSLV-132 or a placebo 13 times over 22 weeks Visit the clinic once every week for the first 2 weeks, then every 2 weeks until the end of treatment and then for a final time 4 weeks later (Day 211) for check-ups, tests and to answer questionnaires about their symptoms Record their symptoms every day on an electronic device

ELIGIBILITY:
Inclusion Criteria:

* Providing written informed consent
* Weight at least 45 kg
* Meet the 2016 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) Classification Criteria for pSS
* Diagnosis in the last 30 years
* Positive anti-Ro/SSA antibody test
* Score of 5 or higher on the EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) scale and the ESSPRI fatigue scale
* Of non childbearing potential or of childbearing potential and using highly effective contraceptive measures

Exclusion Criteria:

* Diagnosis of any active autoimmune disease other than pSS that could affect the efficacy assessments
* Uncontrolled hypothyroidism or severe fibromyalgia
* New medications or change in medications in the last 4 weeks for pSS symptoms
* Receipt of other prohibited medications
* Apheresis or blood donation
* Allergic reaction to RSLV-132 or biologic therapy
* Clinically significant infection in last 30 days
* Participation in another clinical study
* Malignancy in last 5 years
* Positive test for HIV or hepatitis
* Major surgery in last 30 days or anticipated surgery during the study
* Pregnancy or breast feeding
* Laboratory blood tests outside of specified ranges
* Other medical conditions or medications that would make the participant unsuitable

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of cardinal symptoms of Sjogren's | Measured daily from at least 7 days prior to first dose until 169 days after the first dose
  Change from baseline in Sjogren's symptoms on Day 169 assessed using the Sjogren's Symptom Activity Patient Reported Outcome (SSA-PRO) instrument

SECONDARY OUTCOMES:
Tiredness/fatigue assessment | Measured from before the first dose until Day 169
  Change from baseline in the Patient Reported Outcomes Measurement Information System Fatigue Short Form 10a (PROMIS SF10a) on Day 169
RSLV-132 pharmacokinetics | Measured from before the first dose until Day 211
  Serum concentrations of RSLV-132 using an assay measuring RNAse enzyme activity
RSLV-132 immunogenicity | Measured from before the first dose until Day 211
  Presence of antibodies to RSLV-132 measured using an immunoassay
Adverse events | From the first dose of Investigational Product until Day 211
  Incidence of serious and non-serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: James Posada, Study Director — Resolve Therapeutics LLC
Locations (24):
- United States (24):
  - Resolve Clinical Site, Chula Vista, California
  - Resolve Clinical Site, Tustin, California
  - Resolve Clinical Site, Boca Raton, Florida
  - Resolve Clinical Site, Boynton Beach, Florida
  - Evolution Research Center, Hialeah, Florida
  - GNP Research, Hollywood, Florida
  - Resolve Clinical Site, Miami, Florida
  - Life Medical Research, Miami Gardens, Florida
  - Resolve Clinical Site, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Tufts College, Boston, Massachusetts
  - Resolve Clinical Site, Albuquerque, New Mexico
  - Joint and Muscle Research Institute, Charlotte, North Carolina
  - Arthritis and Osteoporosis Consultants of the Carolinas, Charlotte, North Carolina
  - Onsite Clinical Solutions, Salisbury, North Carolina
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Resolve Clinical Site, Nashville, Tennessee
  - Resolve Clinical Site, Austin, Texas
  - Resolve Clinical Site, Katy, Texas
  - Resolve Clinical Site, McKinney, Texas
  - Accurate Clinical Research, Richmond, Texas
  - Resolve Clinical Site, San Antonio, Texas
  - Metrodora Institute, Salt Lake City, Utah
  - Arthritis Northwest, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Posada J, Valadkhan S, Burge D, Davies K, Tarn J, Casement J, Jobling K, Gallagher P, Wilson D, Barone F, Fisher BA, Ng WF. Improvement of Severe Fatigue Following Nuclease Therapy in Patients With Primary Sjogren's Syndrome: A Randomized Clinical Trial. Arthritis Rheumatol. 2021 Jan;73(1):143-150. doi: 10.1002/art.41489. Epub 2020 Nov 22. PMID 32798283
- [Background] Shiboski CH, Shiboski SC, Seror R, Criswell LA, Labetoulle M, Lietman TM, Rasmussen A, Scofield H, Vitali C, Bowman SJ, Mariette X; International Sjogren's Syndrome Criteria Working Group. 2016 American College of Rheumatology/European League Against Rheumatism Classification Criteria for Primary Sjogren's Syndrome: A Consensus and Data-Driven Methodology Involving Three International Patient Cohorts. Arthritis Rheumatol. 2017 Jan;69(1):35-45. doi: 10.1002/art.39859. Epub 2016 Oct 26. PMID 27785888
- See also: Related Info — https://app.patientwing.com/campaign/clinicaltrials.gov